CLINICAL TRIAL: NCT00580203
Title: Collection of Tissue, Blood, and Other Specimens From Patients With Head and Neck Diseases to Study the Causes, Diagnosis, Prevention and Treatment of Cancers
Brief Title: Collection Of Tissue, Blood, and Other Specimens From Patients With Head and Neck Tumors To Study the Causes, Diagnosis, Prevention and Treatment of Cancers
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 04-017
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Cancers
Keywords: HEENT cancers; larynx; thyroid; sarcoma; specimen analysis
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Diseases; Thyroid Diseases; Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and peripheral blood

GROUPS / COHORTS (1):
- 1: Patients with head and neck cancers

SUMMARY:
This is a protocol to collect tissues, blood, and other specimens from patients with malignant or nonmalignant diseases of the head and neck. Collected specimens will be used in laboratory studies to investigate the growth, development, and transformation of normal and abnormal cells in the future.

DETAILED DESCRIPTION:
This is a protocol to collect tissues, blood, and other specimens from patients with malignant or nonmalignant diseases of the head and neck. Collected specimens will be used in laboratory studies to investigate the growth, development, and transformation of normal and abnormal cells in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck diseases are eligible if they have had tissue, serum, urine, or other specimens removed or collected for diagnostic or therapeutic purposes.
* Patients will be entered onto this protocol without preference for any racial or ethnic group.
* Patients may have received prior chemotherapy, radiation, surgical therapy, immunotherapy, or differentiation therapy.
* The specimen collected must be large enough to allow conventional testing necessary for patient care, with the portion of the specimen reserved for research laboratory analysis excised from residual tissue that would otherwise have been discarded.

Exclusion Criteria:

* Patients not giving informed consent will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with head and neck diseases who have had tissue, serum, urine, or other specimens removed or collected for diagnostic or therapeutic purposes.
Sampling Method: Non-Probability Sample
Enrollment: 1468 (Actual)
Dates: Start 2004-02 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Collect tissues, blood, and other specimens from patients with malignant or nonmalignant diseases of the head and neck. Specimens will be used to investigate growth, development, and transformation of normal and abnormal cells in the future. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bhuvanesh Singh, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org